CLINICAL TRIAL: NCT05812859
Title: Novel Vaginal Orthosis for Post-Surgical Healing After Vaginal Reconstructive Surgery For Pelvic Organ Prolapse (NOVa Study)
Brief Title: Vaginal Orthosis Use After Vaginal Reconstructive Surgery
Acronym: NOVa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Max Cadena, Clinical Instructor Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300010943
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Examiner in the post-operative setting will be blinded to intervention during examination and survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Device Use (Experimental): Patient's will use vaginal orthosis daily from the start of week 2 post-operative to week 12 post-operative.
  Interventions: Device: Vaginal Orthosis (COSM Medical)
- Standard of Care (No Intervention): Patient's will proceed with normal standard of care post-operative management which is pelvic rest and light acitvity.

INTERVENTIONS:
Device: Vaginal Orthosis (COSM Medical) — A vaginal orthosis will be 3-D printed by COSM Medical and provided for patients to use from week 2 through week 12 post-operatively. Device will be placed in morning and removed before bed daily.
  Arms: Device Use

SUMMARY:
A novel vaginal orthosis, or splint, made of silicone will be used daily to help support the healing vaginal reconstruction during the post-operative phase from week 2 to week 12.

DETAILED DESCRIPTION:
Background/Rationale:

Pelvic Organ Prolapse (POP) is the bulging or herniation of one or more pelvic organs into or out of the vagina. A woman's estimated lifetime risk of POP is 30-50%, with 2-4% of women being symptomatic. Approximately 300,000 women undergo surgical procedures in the United States to repair POP every year. Recurrence rates of POP after native tissue repair utilizing Sacrospinous Ligament Fixation (SSLF) or Uterosacral Ligament Suspension (USLS) vary based on the definition of surgical or anatomic failure used, however a large RCT reports rate of reoperation at 5 years of 8-11.9%.

With the use of the sacrospinous or uterosacral ligaments for apical support, the long axis of the vaginal canal is deflected posteriorly in the pelvis leaving the anterior wall of the vagina vulnerable to receive more of the downward forces produced intra-abdominally during activity and with absolute increases in intra-abdominal pressure. Given this fact, it is not a coincidence that the area of highest recurrence occurs, despite which definition is used, in the anterior vaginal compartment.

Currently, the standard of care for post-operative management in patients who have undergone native tissue pelvic reconstructive surgery is pelvic rest and reduced activity. The Voices for Pelvic Floor Disorders (Voices PFD) in conjunction with the American Urogynecology Society (AUGS) recommend pelvic rest for a minimum of 6 weeks and for activity to "be up and around, but not too active" for the first two weeks, but to increase ambulation and activity as able with guidance from primary surgeon. By the 6-week post-operative visit, most patients are ready to begin to return to normal daily activities, but some may take a longer time-period of reduced activity.

The "wound" healing process following vaginal surgery starts immediately after hemostasis is achieved and the surgery is completed. The first stage is the inflammatory stage, which has rapid onset and reaches maximal reaction within 1-3 days of surgery. This stage is driven by migration of neutrophils and macrophages responding to factors released from the wound site which are responsible for removal of debris and bacteria in order to prepare the site for the second stage of healing, the proliferative stage. The aim of the proliferative stage is to diminish the surgical site tissue area by contraction and fibroplasia, establishing a viable epithelial barrier to activate keratinocytes. This stage is responsible for the closure of the lesion itself, which includes angiogenesis, fibroplasia, and re-epithelialization. These processes begin in the microenvironment of the lesion within the first 48 hours and can unfold up to the 14th day after the onset of the lesion. With the re-epithelization initiated and Type III collagen now deposited, the remodeling stage or wound maturation begins. The ultimate goal of this third and final stage is to restore or achieve the maximal tensile strength of the healing tissue. This is achieved mainly through the degradation of Type III collagen and production of Type 1 collagen.

The objective of this project is to investigate whether patients who have undergone native tissue pelvic reconstructive surgery for POP would benefit from a supportive intravaginal orthotic device. Participants will be fitted for the device at 2 weeks after surgery with daily use continuing until 12 weeks after surgery, thus providing stabilization during the subepithelial wound healing process leading to improved tissue durability and viability along the repaired vaginal walls.

ELIGIBILITY:
Inclusion Criteria:

1. POP-Q stage 2 to 4 pelvic organ prolapse
2. Vaginal bulge symptoms as indicated by an affirmative response to either question 4 or 5 of the PFDI:

   1. Do you usually have a sensation of bulging or protrusion from the vaginal area?
   2. Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?
3. Undergoing reconstructive vaginal surgery for POP-Q stage 2 to 4 pelvic organ prolapse that must include anterior compartment repair and apical suspension.
4. Willing and able to use and self-manage novel vaginal orthosis after POP surgery from 2 weeks post-operative to 12 weeks post-operative.
5. Available for 2 and 6 weeks, 3, 6, and 12 months follow-up.
6. Able to complete study assessments, per clinician judgement.
7. Able and willing to provide written informed consent.

Exclusion Criteria:

1. Contraindication to surgical intervention as planned in the opinion of the treating surgeon (ie undergoing obliterative procedure).
2. History of previous vaginal reconstructive surgery with or without hysterectomy for POP.
3. Allergy to silicone used in Novel Vaginal Orthosis.
4. Allergy or contraindication to low-dose vaginal estrogen use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective recurrent anterior prolapse | 12 months.
  Pelvic exam will be performed at 12 months post-operative visit and POP-Q measurements will be performed. The "Ba" measurement will be used as the primary outcome comparing the measurements of the vaginal orthosis group and the standard of care group.

SECONDARY OUTCOMES:
Subjective recurrent prolapse | 12 months
  POPDI-6 score will be collected as a part of the PFDI-20 before surgery as well as 3 months, 6 months and 12 months after surgical intervention and change will be compared between groups
Objective recurrent prolapse | 3, 6, and 12 months
  Other measurements of POP-Q system will be compared between groups
Device use complications | 12 months
  Post-operative complications and adverse events will be compared between groups

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No